CLINICAL TRIAL: NCT03346343
Title: Pulmonary Function Using Non-invasive Forced Oscillometry Respiratory Testing: A Prospective Observational Study
Brief Title: Pulmonary Function Using Non-invasive Forced Oscillometry
Acronym: PUFFOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300000296; K23HL157618 (NIH)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Infant, Premature, Diseases; Infant, Newborn, Diseases; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome, Newborn; Meconium Aspiration Syndrome; Transient Tachypnea of the Newborn
MeSH Terms: conditions — Infant, Premature, Diseases; Infant, Newborn, Diseases; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome, Newborn; Meconium Aspiration Syndrome; Transient Tachypnea of the Newborn

STUDY DESIGN:
Intervention Model Description: This will be a single center prospective observational study with pre-specified Aims and Hypotheses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-invasive forced airway oscillometry (Experimental): Analyze lung function using forced airway oscillometry in preterm infants and term infants with and without lung disease with both cross-sectional and longitudinal comparisons.
  Aim 1: Lung function in term and preterm infants without lung disease (anticipated n=264) Aim 2: Lung function in preterm infants with respiratory distress syndrome (RDS) who develop bronchopulmonary dysplasia (BPD) and preterm infants with RDS who do not develop BPD (anticipated n=264) Aim 3: Lung function measurements in infants with common neonatal lung diseases (including RDS, BPD, meconium aspiration syndrome, and transient tachypnea of the newborn) and controls without lung disease (anticipated n=570) Aim 4: Lung function in infants with lung disease before and after common therapeutic interventions
  Interventions: Device: Non-invasive forced airway oscillometry

INTERVENTIONS:
Device: Non-invasive forced airway oscillometry — This is a non-invasive device will measure lung function in spontaneously breathing infants. Infants will have a cushioned mask placed on his/her face and the device will take measurements as the infant breathes normally.

SUMMARY:
The purpose of this observational study is to measure pulmonary function in term and preterm infants with and without pulmonary disease including respiratory distress syndrome, bronchopulmonary dysplasia, transient tachypnea of the newborn, meconium aspiration syndrome, and response to treatments given to newborn infants with lung diseases using a non-invasive airway oscillometry system.

DETAILED DESCRIPTION:
TremoFlo™ N-100 (For Investigational Use Only) Airwave Oscillometry System™ (THORASYS Thoracic Medical Systems Inc. Montreal, Quebec, Canada) is a technology for measuring lung mechanics without patient effort. Pulmonary function testing using flow-volume and lung volumes is one of the most widely used tests to objectively measure lung function in adults. Such measurements are dependent on effort and coordination by the patient which is not possible for newborn infants. The minimum age for spirometry is typically 6 years to master the technique. Therefore, newborn infants usually require forced exhalation, flow interruption, and often sedation/anesthesia in order to obtain accurate pulmonary function measurements. Infant pulmonary function testing can be time-consuming and expensive to perform in newborn infants. This has limited the utilization of this potentially informative method of studying lung function. Measurements of lung function will be particularly informative during transition from having lungs filled with fluid during intra-uterine life to having lungs filled with air in extra-uterine life in preterm and term babies without lung disease, as well as in newborn infants with lung diseases including respiratory distress syndrome, bronchopulmonary dysplasia, transient tachypnea of the newborn, meconium aspiration syndrome, and after the effects of treatments given to newborn infants with lung diseases.

The TremoFlo device uses the forced oscillation technique during spontaneous infant breathing and notably does not require any sedation to perform. The forced oscillation technique measures lung function by superimposing a gentle multi-frequency airwave onto the infant's respiratory airflow while the infant breathes spontaneously. Only a short period of breathing is required to obtain a reliable measurement of airway resistance and reactance. Oscillometry has been successfully utilized to quantify lung function in asthmatic children and adults with chronic obstructive pulmonary disease, but never previously in infants. This proposal brings this non-invasive technique of measuring lung function to the neonatal population to identify changes in respiratory mechanics between term and pre-term gestations and quantify fluctuations in infant lung function in response to disease progression and therapeutic intervention. The ease of oscillometry that only requires tidal breathing eliminates the need for patient cooperation and maneuvers that previously excluded lung function testing in the neonatal intensive care unit. This proposal will evaluate the feasibility and clinical value of oscillometry in newborns, both to detect changes in premature compared to full-term gestations as well as disease cohorts by introducing functional measures of lung function to bedside care.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age at least 22 weeks at birth
* Infants off ventilator/continuous positive airway pressure ≥ 12 hours
* Infants whose parents/legal guardians have provided consent

Exclusion Criteria:

* Infants with major malformation
* Infants with a neuromuscular condition that affects respiration
* Infants with terminal illness
* Infants with a decision made to withhold or limit support

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klinger AP, Travers CP, Martin A, Kuo HC, Alishlash AS, Harris WT, Carlo WA, Ambalavanan N. Non-invasive forced oscillometry to quantify respiratory mechanics in term neonates. Pediatr Res. 2020 Aug;88(2):293-299. doi: 10.1038/s41390-020-0751-7. Epub 2020 Jan 14. PMID 31935746

RESULTS

PARTICIPANT FLOW:
Groups:
- Bronchopulmonary Dysplasia at 36 Weeks: Infants with a diagnosis of bronchopulmonary dysplasia based on respiratory support at 36 weeks' postmenstrual age
- Infant Respiratory Distress Syndrome: Infants with a diagnosis of respiratory distress syndrome based on initial requirement for respiratory support but who did not meet criteria for BPD
- Preterm no RDS/BPD: Preterm infants with no RDS or BPD
- Control: Term/Late Preterm infants with no respiratory disease
Period: Overall Study
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
Started | 133 | 228 | 94 | 145
Completed | 133 | 228 | 94 | 145
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control | Total
Number analyzed (Participants) | 133 | 228 | 94 | 145 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 133 | 228 | 94 | 145 | 600
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 121 | 50 | 72 | 311
  Male | 65 | 107 | 44 | 73 | 289
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 4 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 77 | 90 | 42 | 46 | 255
  White | 56 | 133 | 48 | 93 | 330
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 3 | 5 | 24
  Not Hispanic or Latino | 127 | 218 | 91 | 140 | 576
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Gestational Age [Mean (Standard Deviation); unit: weeks] — Gestational age at birth in weeks
  weeks | 25 (2) | 29 (3) | 33 (2) | 38 (1) | 31 (2)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Reactance Curve (AXR)
Description: AXR as the measure of overall measure of reactance of the respiratory system quantified by oscillometry and measured in cmH2O/L
Time Frame: 40 weeks' postmenstrual age or discharge until 2 years
Measure: Mean (Standard Deviation); unit: cmH2O/L
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
Number analyzed (Participants) | 123 | 221 | 93 | 145
cmH2O/L | 733 (257) | 599 (212) | 495 (159) | 385 (198)

2. Secondary Outcome: R7-20
Description: Difference between resistance at 7 Hz and 20 Hz in the respiratory system quantified by oscillometry and measured in cmH2O·s/L
Time Frame: 40 weeks' postmenstrual age or discharge until 2 years
Measure: Mean (Standard Deviation); unit: cmH2O·s/L
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
Number analyzed (Participants) | 123 | 221 | 93 | 145
cmH2O·s/L | 24 (10) | 20 (8) | 17 (6) | 13 (9)

3. Secondary Outcome: R7
Description: Resistance at 7 Hz in the respiratory system quantified by oscillometry and measured in cmH2O·s/L
Time Frame: 40 weeks' postmenstrual age or discharge until 2 years
Measure: Mean (Standard Deviation); unit: cmH2O·s/L
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
Number analyzed (Participants) | 123 | 221 | 93 | 145
cmH2O·s/L | 56 (16) | 51 (13) | 46 (9) | 40 (13)

4. Secondary Outcome: X7
Description: Reactance at 7 Hz in the respiratory system quantified by oscillometry and measured in cmH2O·s/L
Time Frame: 40 weeks' postmenstrual age or discharge until 2 years
Measure: Mean (Standard Deviation); unit: cmH2O·s/L
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
Number analyzed (Participants) | 123 | 221 | 93 | 145
cmH2O·s/L | -53 (21) | -45 (16) | -39 (10) | -34 (13)

5. Secondary Outcome: Longer-term Pulmonary Outcomes
Description: Severe morbidity: respiratory support including or CPAP or ventilation or tracheostomy; moderate morbidity: supplemental oxygen; treatment with daily pulmonary medications; ≥2 rehospitalizations for respiratory illness; ≥3 episodes of wheeze ≥2 weeks apart; mild morbidity: treatment with intermittent pulmonary medications; ≥2 episodes of wheeze ≥2 weeks apart; ≥2 medical visits for respiratory illness ≥2 weeks apart; 1 rehospitalization for respiratory illness)
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-10

ADVERSE EVENTS:
Time Frame: During oscillometry testing from beginning of test until completion of test up to 30 minutes
Description: Desaturations or bradycardia events during oscillometry testing
Arm/Group | Bronchopulmonary Dysplasia at 36 Weeks | Infant Respiratory Distress Syndrome | Preterm no RDS/BPD | Control
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/228 | 0/94 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/228 | 0/94 | 0/145
Other Adverse Events (participants affected / at risk) | 0/133 | 0/228 | 0/94 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03346343/Prot_SAP_000.pdf